CLINICAL TRIAL: NCT07336758
Title: A Human Absorption, Distribution, Metabolism and Excretion (hADME) and Absolute Bioavailability Trial After a Single Micro-tracer Dose of BI 1584862 (C-14) and a Single, Concomitant, Intravenous Micro-dose of BI 1584862 (C-13) in Healthy Male Trial Participants (a Phase I, Open-label, Non-randomised, Single-dose, Fixed-sequence Trial)
Brief Title: A Study in Healthy Men to Test How BI 1584862 is Processed in the Body
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1484-0017; 2025-522311-41-00 (Registry Identifier: CTIS); U1111-1322-4722 (Registry Identifier: WHO Registry)
Record Dates: First submitted 2026-01-02; First posted 2026-01-13 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BI 1584862 (C-14) (Test treatment) followed by [13C]-labeled BI 1584862 (Reference treatment) (Experimental)
  Interventions: Drug: [13C]-labeled BI 1584862; Drug: Unlabeled BI 1584862 mixed with [14C]-labeled BI 1584862

INTERVENTIONS:
Drug: [13C]-labeled BI 1584862 — [13C]-labeled BI 1584862, Reference treatment
Drug: Unlabeled BI 1584862 mixed with [14C]-labeled BI 1584862 — BI 1584862 (C-14), Test treatment

SUMMARY:
The goal of this study is to find out how BI 1584862 moves through and exits the body of healthy men. To do this, BI 1584862 is labelled using radioactive carbon (C-14) and using a non-radioactive, naturally occurring, stable isotope (C-13). The study will measure how much of the study medicine is recovered in urine and faeces after taking it by mouth. It will also look at how much of the study medicine enters the bloodstream when taken by mouth compared to a small dose given directly into the bloodstream. The study staff measures the amount of BI 1584862 and its broken-down parts in the blood, the urine, and the stool.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male trial participant according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
2. Age of 18 to 55 years (inclusive) at screening
3. BMI of 18.5 to 29.9 kg / m2 (inclusive) at screening
4. Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial

Exclusion Criteria:

1. Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
4. Any evidence of a concomitant disease assessed as clinically relevant by the investigator Further exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2026-01-22 (Actual); Primary Completion 2026-03-04 (Estimated); Study Completion 2026-03-04 (Estimated)

PRIMARY OUTCOMES:
Fraction excreted in urine as percentage of the administered dose over the time interval from 0 to the last quantifiable time point (feurine,0-tz) | Up to Day 14
  hADME part
Fraction excreted in faeces as percentage of the administered dose over the time interval from 0 to the last quantifiable time point (fefaeces,0-tz) | Up to Day 14
  hADME part
Sum of feurine,0-tz and fefaeces,0-tz (total recovery of [14C]-radioactivity) | Up to Day 14
  hADME part
Area under the concentration-time curve of the analyte over the time interval from 0 extrapolated to infinity in plasma) of BI 1584862 after a single oral administration of BI 1584862 (C-14) (AUC0-∞) | Up to day 13
  BA part
Area under the concentration-time curve of the analyte over the time interval from 0 extrapolated to infinity in plasma) of [13C]-BI 1584862 after a single intravenous infusion of BI 1584862 (C-13) (AUC0-∞) | Up to Day 6
  BA part

SECONDARY OUTCOMES:
Cmax (maximum measured concentration of the analyte in plasma) of BI 1584862 after a single oral administration of BI 1584862 (C-14) | Up to Day 13
  hADME and BA part
AUC0-tz (area under the concentration-time curve of the analyte over the time interval from 0 to the last quantifiable time point in plasma) of BI 1584862 after a single oral administration of BI 1584862 (C-14) | Up to Day 13
  hADME and BA part
Cmax of [14C]-radioactivity after a single oral administration of BI 1584862 (C-14) | Up to Day 13
  hADME part
AUC0-tz of [14C]-radioactivity after a single oral administration of BI 1584862 (C-14) | Up to Day 13
  hADME part
Cmax of [13C]-BI 1584862 after a single intravenous administration of BI 1584862 (C-13) | Up to Day 6
  BA part
AUC0-tz of [13C]-BI 1584862 after a single intravenous administration of BI 1584862 (C-13) | Up to Day 6
  BA part

CONTACTS AND LOCATIONS:
Locations (1):
- ICON-Groningen-62040, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization). For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com